CLINICAL TRIAL: NCT04784689
Title: Host Immune Response to Novel RNA COVID-19 Vaccination in Patients With Cancer (CTMS# 21-0012)
Brief Title: Host Immune Response to Novel RNA COVID-19 Vaccination
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Kate Lathrop, Clinical Investigator, The University of Texas Health Science Center at San Antonio
Other Study IDs: CTMS 21-0012
Record Dates: First submitted 2021-03-03; First posted 2021-03-05 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: COVID-19 Vaccine; Cancer
MeSH Terms: conditions — Neoplasms | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective - Cancer Patients that have received COVID-19 Vaccination
  Interventions: Biological: COVID-19 Vaccine

INTERVENTIONS:
Biological: COVID-19 Vaccine — COVID-19 Vaccine

SUMMARY:
To determine the antibody response level in patients with cancer to the COVID-19 vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Must be eligible to receive the COVID19 vaccination by standard and current CDC guidelines. This includes all RNA vaccinations grant EUA status by the FDA
3. Diagnosed with any malignancy within the last 5 years, with the exception of early-stage squamous cell skin cancer, early-stage basal cell skin carcinoma and noninvasive pathology such as DCIS (Ductal Carcinoma in-situ)
4. Able to provide informed consent
5. Patients can be on any form of treatment (including clinical trials) and at any stage (including remission) in their cancer therapy plan - including chemotherapy, immunotherapy, targeted therapy, hormonal therapy, radiation, palliative care or observation.

Exclusion Criteria:

1. Previously documented COVID infection
2. Previously enrolled in a vaccination trial and either still blinded or known to receive the vaccination. (Those patients on a trial but known to receive a placebo dose are eligible to enroll)
3. Contraindication to the vaccination based on current CDC guideline such as know allergic reactions that increase risk of having an allergic reaction to a COVID RNA vaccination. This includes but is not limited to:

   * Severe allergic reaction (e.g., anaphylaxis) after a previous dose of an mRNA COVID-19 vaccine or any of its components
   * Immediate allergic reaction of any severity to a previous dose of an mRNA COVID-19 vaccine or any of its components (including polyethylene glycol [PEG])
   * Immediate allergic reaction of any severity to polysorbate (due to potential cross-reactive hypersensitivity with the vaccine ingredient PEG)
4. Pregnant or breastfeeding
5. Unable to comply with study related procedures as determined by the study team.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Mays Cancer Center patients eligible to receive the COVID-19 vaccination.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-05-18 (Actual)

PRIMARY OUTCOMES:
Antibody response level in patients with cancer to the COVID-19 vaccination. | Pre dose on day 1 (baseline), pre dose on day 21, day 35, 6 months, 12 month and 18 months
  Antibody response change over time

CONTACTS AND LOCATIONS:
Overall Officials: Dimpy Shah, MD PhD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- Mays Cancer Center, UT Health San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided